CLINICAL TRIAL: NCT06802211
Title: The Effect of Discontinuing Estrogen Containing Oral Contraceptives on Corticosteroid-binding Globulin and Total Cortisol Concentrations
Brief Title: CBG Normalization After Discontinuation of COC's
Status: Not yet recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Annemieke Heijboer, Prof. Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL87932.018.24
Record Dates: First submitted 2025-01-24; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Cessation of Combined Oral Contraceptive Use
Keywords: CBG; corticosteroid-binding globulin; total cortisol; combined oral contraceptives; COCs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In this study, the investigators aim to examine after which duration corticosteroid-binding globulin (CBG) and total cortisol concentrations return to normal after cessation of the combined oral contraceptive pill in healthy women.

DETAILED DESCRIPTION:
Use of exogenous estrogens is known to increase corticosteroid-binding globulin (CBG) levels and thereby total cortisol concentrations measured in serum. When endocrine function are performed to assess hypothalamus-pituitary-adrenal function, total cortisol levels are measured in serum. When women use exogenous oral estrogen, for instance the birth control pill, the current recommendation is to discontinue oral estrogens for at least 6 weeks before the test. This may introduce diagnostic delay and inconvenience for the patient. The duration it takes for CBG concentrations to return to normal, have not been studied in vivo as far as known by the investigators.

The main objective of this prospective observational study is to determine the duration in which CBG and total cortisol concentrations return to normal after cessation of oral estrogen. Secondary objectives are to examine the normalization of other hormone binding proteins and their corresponding hormones (VDBP & vitamin D; TBG & T4, T3; SHBG & testosterone; IGFBP3 & IGF1).

The study population consists of healthy women aged ≥18 years old, who are planning to stop using combined oral contraceptives (COCs) for at least six weeks. The study consists of 8 weekly blood samples. The first blood sample will be performed one week before cessation of COCs, the second one at the moment of cessation and after cessation the next six weekly blood samples will be taken.

After establishing when values return to normal, doctors have a better idea of how many weeks after stopping COCs, blood results can be properly assessed. If the duration were shorter than six weeks, this would mean less inconvenience for women undergoing dynamic function tests who would have to stop taking their contraceptive pill.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Using oral combined contraceptives of any kind and dosage
* Planning to stop COC use shortly for at least 6 weeks (out of own reasons such as a pregnancy wish or choice for non-hormone based contraceptives)
* COC use for at least 3 consecutive weeks before the discontinuation
* Ability to provide informed consent
* Ability to speak and understand Dutch

Exclusion Criteria:

* Switching to other hormonal contraceptives after taking the COC pill (e.g. progesterone containing contraceptives such as the Mirena IUD, contraceptive implants) directly after the discontinuations
* Contra-indications to quit COC
* Biological factors that affect CBG concentrations, including:

  * Illnesses interfering with CBG levels (severe liver or kidney disease, active malignancy, hyperthyroidism)
  * Use of insulin, systemic exogenous glucocorticoids, mitotane, selective estrogen receptor modulators (SERMs)
  * Pregnancy during study period after discontinuation of COCs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult females who are planning to discontinue estrogen containing oral contraceptives for a duration of at least 6 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Time to normalization of CBG and total cortisol concentrations | 8 weeks
  Time in weeks until plateau is reached.

SECONDARY OUTCOMES:
Time to normalization of VDBP, vitamin D, TBG, T4, T3, SHBG, testosterone, IGFBP3 and IGF1 | 8 weeks
  Time in weeks until plateau is reached.

OTHER OUTCOMES:
Estradiol concentration | 8 weeks
  Used for determining menstrual cycle
Progesterone concentration | 8 weeks
  Used for determining menstrual cycle
LH concentration | 8 weeks
  Used for determining menstrual cycle
FSH concentration | 8 weeks
  Used for determining menstrual cycle
Occurrence of vaginal blood loss | 8 weeks
  Used for determining menstrual cycle
Albumin concentration | 8 weeks
Prolactin concentration | 8 weeks
fT3 and fT4 concentration | 8 weeks
TSH concentration | 8 weeks
HCG concentration | Measured at 6th week after cessation of COCs

CONTACTS AND LOCATIONS:
Overall Officials: Annemieke C Heijboer, Prof. Dr., Principal Investigator — Amsterdam UMC location Vrije Universiteit Amsterdam, Department of Laboratory Medicine, Endocrine Laboratory, Boelelaan 1117, Amsterdam, The Netherlands

IPD SHARING:
Plan to Share IPD: No